CLINICAL TRIAL: NCT05772663
Title: Elaboration and Evaluation of a Program of Self-rehabilitation Based on Daily Living Activities in Patients With Chronic Stroke
Brief Title: A Rehabilitation Program Based on Daily Activities in Patients With Cerebrovascular Accident
Acronym: LARAQS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: APHP220833; 2023-A00302-43 (Registry Identifier: IDRCB)
Record Dates: First submitted 2023-02-10; First posted 2023-03-16 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-09

CONDITIONS: Stroke
Keywords: Stroke; self-rehabilitation program
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- personalized program group (Experimental): people with chronic stroke
  Interventions: Other: Personalized program of rehabilitation
- routine rehabilitation care group (Active Comparator): people with chronic stroke
  Interventions: Other: Routine program of rehabilitation

INTERVENTIONS:
Other: Personalized program of rehabilitation — D56: Follow-up visit (D56). Assessments: AMPS, MCRO, Satisfaction VAS. Installation of accelerometer wristbands for the sub-sample of 40 people with stroke drawn at random secondary accelerometry analysis.
  Between D56 and D112: For 8 weeks, the person does not receive any intervention apart from their usual rehabilitation. At D63, the person returns the accelerometric wristbands.
  D112: The assessments carried out by occupational therapist are: AMPS, MCRO. Installation of accelerometer bracelets for the sub-sample of 40 people with stroke, randomly selected for secondary analysis on accelerometers (subjects from the two groups, experimental and control, i.e. 20*20). At D119, the person returns the accelerometric writbands.
  Arms: personalized program group
Other: Routine program of rehabilitation — Assessments: AMPS, MCRO, Satisfaction VAS. Installation of accelerometer wristbands for the sub-sample of 40 people with stroke drawn at random secondary accelerometry analysis.
  Between D56 and D112: For 8 weeks, the person does not receive any intervention apart from their usual rehabilitation. At D63, the person returns the accelerometric wristbands.
  D112: The assessments carried out by occupational therapist are: AMPS, MCRO. Installation of accelerometer bracelets for the sub-sample of 40 people with stroke, randomly selected for secondary analysis on accelerometers (subjects from the two groups, experimental and control, i.e. 20*20). At D119, the person returns the accelerometric writbands.
  Arms: routine rehabilitation care group

SUMMARY:
Mixed qualitative and quantitative study, in two phases:

Creation of a self-rehabilitation program based on people's daily living activities and designed with and for them.

Randomized controlled study to explore whether there is a potential benefit for patients with chronic stroke to use a self-rehabilitation program.

DETAILED DESCRIPTION:
In France, stroke affects nearly 150,000 people per year and is therefore a major problem public health in France but also in Europe . With improved support treatment, the mortality rate decreases, but the sequelae, linked to the consequences of the stroke, remain numerous . More than 88% of stroke victims return at home upon discharge from hospital rehabilitation. However more and more people experience difficulties as a result of this return. Hospital discharge entails an imbalance between the period of hospitalization and place of residence in terms of the frequency and intensity of rehabilitation. In fact, the person benefits from rehabilitation during his hospitalization daily. After returning home, the person no longer benefits only 1 to 2 rehabilitation sessions per week, sometimes less . In view of these different elements, the investigators issue the assumption that making available to people AVC a self-rehabilitation program designed with and for them and centered on the meaningful occupations of the person will allow an increase in their occupational performance in their life activities daily. The aim of this study is to create a self-rehabilitation program based on people's daily living activities and designed with and for them and to evaluate the benefits of this program with a randomized controlled study.

ELIGIBILITY:
Inclusion Criteria:

* Having had a stroke ischemic or hemorrhagic for more than 6 months before inclusion in the study.
* Having had a single cerebral hemispheric lesion
* Patient informed and having signed consent

Exclusion Criteria:

-Patient under guardianship or curatorship

* Pregnant or breastfeeding women
* Cognitive impairment defined by BDAE <3
* Previous operation of the paretic limb at course of the last 6 months at inclusion
* Total absence of motor skills in the upper limb hemiplegic

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2028-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Assessment of Motor and Process Skills AMPS° | Day -7
  The Assessment of Motor and Process Skills (AMPS) is an observational assessment that allows for the simultaneous evaluation of motor and process skills and their effect on the ability of an individual to perform complex or instrumental and personal activities of daily living (ADL). The AMPS is comprised of 16 motor and 20 process skill items.
Assessment of Motor and Process Skills AMPS° | Day 0
  The Assessment of Motor and Process Skills (AMPS) is an observational assessment that allows for the simultaneous evaluation of motor and process skills and their effect on the ability of an individual to perform complex or instrumental and personal activities of daily living (ADL). The AMPS is comprised of 16 motor and 20 process skill items.
Assessment of Motor and Process Skills AMPS° | Day 56
  The Assessment of Motor and Process Skills (AMPS) is an observational assessment that allows for the simultaneous evaluation of motor and process skills and their effect on the ability of an individual to perform complex or instrumental and personal activities of daily living (ADL). The AMPS is comprised of 16 motor and 20 process skill items.
Assessment of Motor and Process Skills AMPS° | Day112
  The Assessment of Motor and Process Skills (AMPS) is an observational assessment that allows for the simultaneous evaluation of motor and process skills and their effect on the ability of an individual to perform complex or instrumental and personal activities of daily living (ADL). The AMPS is comprised of 16 motor and 20 process skill items.

SECONDARY OUTCOMES:
Canadian Occupational Performance Measure (COPM) | Day -7
  The Canadian Occupational Performance Measure is an evidence-based outcome measure designed to capture a client's self-perception of performance in everyday living, over time.
Canadian Occupational Performance Measure (COPM) | Day 0
  The Canadian Occupational Performance Measure is an evidence-based outcome measure designed to capture a client's self-perception of performance in everyday living, over time.
Canadian Occupational Performance Measure (COPM) | Day 56
  The Canadian Occupational Performance Measure is an evidence-based outcome measure designed to capture a client's self-perception of performance in everyday living, over time.
Canadian Occupational Performance Measure (COPM) | Day 112
  The Canadian Occupational Performance Measure is an evidence-based outcome measure designed to capture a client's self-perception of performance in everyday living, over time.
Satisfaction. Visual Analogic Scale (Satisfaction VAS) | D56
  To assess post-stroke satisfaction with the program, we will use a Visual Analog Scale (0-10)
program acceptance score | Day 56
  Acceptance questionnaire
program acceptance score | Day 112
  Acceptance questionnaire
Quantity of acceleration (accelerometer wristbands) | Day-7
  Quantity of acceleration per upper limb (number of acceleration) It will be established on the basis of an accelerometer wearing time of 168 hours (7 days continuously).
Quantity of acceleration (accelerometer wristbands) | Day 56
  Quantity of acceleration per upper limb (number of acceleration) It will be established on the basis of an accelerometer wearing time of 168 hours (7 days continuously).
Quantity of acceleration (accelerometer wristbands) | Day 112
  Quantity of acceleration per upper limb (number of acceleration) It will be established on the basis of an accelerometer wearing time of 168 hours (7 days continuously).
Time spent doing the program | at the end of the study, un average of 56 days
  To assess adherence to the self-rehabilitation program, investigators will use a monitoring notebook completed by the person with stroke on the follow-up of sessions / self-rehabilitation time.
  Outcome measure in time (hours per week)

CONTACTS AND LOCATIONS:
Overall Officials: Samuel POUPLIN, PhD, Principal Investigator — New technology Platform department, Raymond Poincaré hospital -APHP
Locations (1):
- New Technilogy Platform department, Raymond Poincaré hospital - APHP, Garches, France

IPD SHARING:
Plan to Share IPD: No